CLINICAL TRIAL: NCT00495976
Title: A Pilot Study to Investigate the Effects of Hot Drinks on Nasal Airway Resistance and Symptoms of Common Cold
Brief Title: Study to Investigate the Effects of Hot Drinks on Nasal Airway Resistance and Symptoms of Common Cold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Professor Ron Eccles, Cardiff University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hot drink
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Common Cold/Flu
Keywords: common cold; flu; influenza
MeSH Terms: conditions — Common Cold; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: A commercially produced cordial drink

SUMMARY:
Common cold medicines are often formulated as a hot drink yet there is no evidence in the public domain that presenting the medicine as a hot drink has any impact on symptom severity.

DETAILED DESCRIPTION:
Common cold medicines are often formulated as a hot drink and usually contain paracetamol and a decongestant such as phenylephrine but it is the 'hot drink' formulation that is often an attraction to the patient in deciding on which formulation of a cold medicine to purchase and use. Hot drinks have been used to relieve the symptoms of acute respiratory infections such as colds and flu for hundreds of years and are found in the traditional medicines of countries throughout the world. The idea of using a hot drink to treat colds and flu appears to originate from a perceived link between exposure to cold and chilling and the onset of a respiratory infection. In order to combat the cold exposure many traditional remedies use a warming and soothing drink or application of a warming ointment . Despite the widespread folklore that hot drinks are an effective treatment for colds and flu, and the use of hot drink formulations for many current common cold medicines, there appears to be no evidence base in the medical literature supporting the efficacy of this common treatment for common cold. The aim of the present study is to obtain new knowledge about the effects of hot drinks on nasal airway resistance and other symptoms of common cold.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years.
* Has given informed consent.
* Is suffering from common cold/flu like illness
* Indicates they are suffering from at least three common cold symptoms (runny nose, sneezing, blocked nose, sore throat, cough) and scores at least 2 symptoms as moderate on four point ordinal scale of (0=not present, 1=mild, 2=moderate, 3=severe)

Exclusion Criteria:

Subjects will not be enrolled in the study if any of the following criteria are met:

* The subject is unwilling to sign the consent form.
* The subject has a clinically significant cardiovascular, endocrinological, neurological, respiratory, gastrointestinal disease or any other disease that is considered by the investigator as a reason for exclusion.
* The subject has a severe nasal septal deviation or other condition that could cause nasal obstruction such as the presence of nasal polyps.
* The subject has had nasal surgery in the past that in the opinion of the investigator may influence symptom scores or nasal airway resistance
* The subject has ingested any alcohol within the previous 12 hours or more than 4 units of alcohol in the previous 24 hours
* The subject is a drug or alcohol abuser
* The subject is taking any prescribed medication other than for contraception
* The subject has had common cold for more than 7 days
* The subject has recently taken a common cold medicine that in the opinion of the investigator may influence symptom scores or nasal airway resistance (analgesics, nasal decongestants, cough medicines)
* The subject has ingested any hot food or drink within the previous hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in nasal conductance of airflow from before the drink to immediately after the drink | prospective

SECONDARY OUTCOMES:
Exploratory analysis will also be made to investigate the relationship between objective measures of nasal airflow and the symptoms of common cold. | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Ron Eccles, D.Sc, Principal Investigator — Common Cold Centre and Healthcare Clinical Trials, Cardiff University, UK
Locations (1):
- Common Cold Centre and Healthcare Clinical Trials, Cardiff, Wales, United Kingdom

REFERENCES:
- [Result] Sanu A, Eccles R. The effects of a hot drink on nasal airflow and symptoms of common cold and flu. Rhinology. 2008 Dec;46(4):271-5. PMID 19145994
- See also: Common Cold Centre Cardiff University UK — http://www.cf.ac.uk/biosi/subsites/cold/
- See also: Healthcare Clinical Trials — http://www.cf.ac.uk/biosi/subsites/cold/trial2.html